CLINICAL TRIAL: NCT03074266
Title: Clinical Performance of the Investigational GEM Hemochron® 100 in Populations Ages 18 Years and Older
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Accriva Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: HRZ-CSS-15-0002
Record Dates: First submitted 2017-03-01; First posted 2017-03-08 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Blood Coagulation Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Blood coagulation test 1: Therapeutic: Waste blood from heparinized patients undergoing interventional procedures (standard of care) in different clinical settings will be used to conduct coagulation tests using GEM Hemochron 100 during the course of the procedure before ("baseline") and after heparin administration.
  There is no drug administration or therapeutic intervention in this study. The interventional procedure (described above) is standard of care and all results of blood coagulation testing using GEM Hemochron 100 performed in this study are not used to influence that care.
  Interventions: Diagnostic Test: GEM Hemochron 100 ACT
- Blood coagulation test 2: Therapeutic: Waste blood from heparinized patients undergoing interventional procedures (standard of care) in different clinical settings will be used to conduct duplicate coagulation tests using Signature Elite during the course of the procedure before ("baseline") and after heparin administration.
  There is no drug administration or therapeutic intervention conducted in the course of this study. The interventional procedure (described above) is standard of care. The only difference in standard of care is that the blood coagulation test is run in duplicate.
  Interventions: Diagnostic Test: GEM Hemochron 100 ACT

INTERVENTIONS:
Diagnostic Test: GEM Hemochron 100 ACT — Activated Clotting Time

SUMMARY:
This study is designed to evaluate and verify the clinical accuracy of the Hemochron® MCS 7000 Whole Blood Microcoagulation System; a point-of-care, whole blood Activated Clotting Time (ACT) measurement in comparison with the Hemochron Signature Elite® Whole Blood Microcoagulation System; a 510(k) cleared predicate device. This is a multi-center, prospective method comparison, with data to be analyzed separately from each site as well as combined for all sites.

DETAILED DESCRIPTION:
The study will be performed in the clinical setting by trained professional operators.

Group 1: Whole Blood Coagulation Test 1, GEM Hemochron® 100

Group 2: Whole Blood Coagulation Test 2, Hemochron® Signature Elite® 7000 Whole Blood Microcoagulation System

Ex-vivo whole blood samples destined for discard after all medically directed tests are complete will be used from heparinized patients undergoing standard of care interventional procedures in different clinical settings. These include, but are not limited to, the cardiovascular operating room (CVOR), cardiac catheterization lab, surgical intensive care unit (SICU), the electrophysiology (EP) lab, and in extracorporeal membrane oxygenation (ECMO) applications.

A distribution of ACT values is necessary to evaluate clinical accuracy. The target number of subjects for each site is 100.

Samples will be examined at baseline (pre-heparin administration) and at the end of the procedure. Heparinized samples may be obtained for ACT testing once or multiple times while heparin is administered throughout the duration of the procedure. The frequency and time intervals of ACT testing will be determined by the Standard of Care. No additional blood volume or extra blood draws will occur as the result of this study.

The work flow for the testing process will be consistent across all sites. Expected duration of the study is dependent upon the site logistics but generally is expected to last no more than four to six weeks.

ACT results generated from the GEM Hemochron 100 instrument during this study will be used solely for research purposes and will not be used for anticoagulation management of study subjects. No patient follow up is required.

The study will include two GEM Hemochron 100 instruments, trained operators, and two Signature Elite instruments for each procedure.

Guidance was obtained from Point-of-Care Monitoring of Anticoagulation Therapy; Approved Guideline (CLSI POCT14-A), CLSI EP09-A3: "Method Procedure Comparison and Bias Estimation Using Patient Samples; Approved guideline Third Edition" and peer reviewed literature.

All study data will be collected on Case Report Forms and all analysis will be performed by Accriva.

ELIGIBILITY:
Inclusion Criteria:

Therapeutic Group

Patients meeting all of the following criteria will be considered for entry into the study:

* Males and females 18 years or older.
* Patients scheduled for elective or urgent procedures requiring anticoagulation with UFH.
* Patients requiring heparin anticoagulant therapy for any approved indication and being managed and monitored with the ACT test.

Exclusion Criteria:

The following criteria define the population of subjects who will not be accepted in the study:

* The subject develops a significant, unexpected, concurrent illness or adverse event before the first whole blood sample is drawn.
* The subject with a hematocrit of less than 20% or greater than 55% since these samples are not recommended for testing due to optical densities outside of the Hemochron instrument levels of detection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population to be studied consists of subjects who require parenteral anticoagulant therapy with UFH in accordance with the approved label indications for heparin administration.
  • Therapeutic Group (T): Patients pre-heparin Patients undergoing procedure requiring anticoagulation with UFH
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Hemochron® MCS 7000 Whole Blood Microcoagulation System ACT measurements (time of whole blood coagulation in seconds) are clinically equivalent to those of the Hemochron Signature Elite® Whole Blood Microcoagulation System | Therapeutic: 1 day; Normal: 1 day (duration of a single venous blood collection)
  Demonstrate that the Hemochron® MCS 7000 Whole Blood Microcoagulation System Activated Clotting Time (ACT) measurements (time of whole blood coagulation in seconds) are clinically equivalent to those of the Hemochron Signature Elite® Whole Blood Microcoagulation System; a 510(k) cleared predicate device

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rubinstein, MD, Study Director — Accriva Diagnostics
Locations (9):
- United States (9):
  - Accriva Study Site, Los Angeles, California
  - Accriva Study Site, Sacramento, California
  - Accriva Study Site, Aurora, Colorado
  - Accriva Study Site, Baltimore, Maryland
  - Accriva Study Site, Takoma Park, Maryland
  - Accriva Study Site, New Brunswick, New Jersey
  - Accriva Study Site, Chapel Hill, North Carolina
  - Accriva Study Site, Falls Church, Virginia
  - Accriva Study Site, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No